CLINICAL TRIAL: NCT04111471
Title: The Use of Inulin to Prevent Dysbiosis in Pediatric Hematopoietic Stem Cell Transplant Recipients
Brief Title: The Use of A Prebiotic to Promote a Healthy Gut Microbiome in Pediatric Stem Cell Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Mehreen Arshad, Fellow of Pediatric Infectious Diseases, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2019-2801
Record Dates: First submitted 2019-06-25; First posted 2019-10-01 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Microbial Colonization
Keywords: Microbiome; Prebiotic
MeSH Terms: conditions — Communicable Diseases | interventions — Prebiotics; Inulin; maltodextrin

STUDY DESIGN:
Intervention Model Description: Qualified patients that are admitted to Lurie Children's Hospital and agree to participate will either be randomized to receive the placebo or prebiotic, inulin. Randomization will occur 1:1
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants will be randomized by an independent statistician based on patient enrollment number (LCH 001- LCH 040). Randomization will be 1:1. The statistician will randomly assort LCH 001-020 into Inulin/Placebo and LCH 021- LCH 040 into Inulin/placebo. This will ensure that an equal number of enrolled participants will be in each arm at 20 patients, and then again at anticipated full 40 patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Arm (Placebo Comparator): 20 patients will receive 5.6 g of placebo product (maltodextrin) daily for a total of 21 days (7 days before and until 2 weeks after transplant)
  Interventions: Dietary Supplement: Placebos
- Prebiotic (Inulin) Arm (Experimental): 20 patients will receive 10 g of inulin product daily for a total of 21 days (7 days before and until 2 weeks after transplant)
  Interventions: Dietary Supplement: Prebiotics

INTERVENTIONS:
Dietary Supplement: Prebiotics — Enrolled patients will receive 10 grams of inulin daily for 21 days
  Other Names: inulin
  Arms: Prebiotic (Inulin) Arm
Dietary Supplement: Placebos — Enrolled patients will receive 5.6 grams of placebo powder daily for 21 days
  Other Names: Maltodextrin
  Arms: Placebo Arm

SUMMARY:
This study will look at the effect of the prebiotic inulin compared to placebo on children undergoing stem cell transplant.

DETAILED DESCRIPTION:
Children enrolled in the study will receive either the prebiotic inulin or a placebo for 21 days during the study period. They will start taking the product seven days before transplant starts until 14 days after transplant. Stool will be collected twice weekly until thirty days after transplant or discharge, whichever occurs first. Stool samples will be sampled for metagenomic sequencing to identify the diversity of bacteria within the stool. They will also be analyzed for amount of short-chain fatty acid content (a breakdown product of inulin) as well as for presence of genes that confer antibiotic resistance. From 30 days after transplant until 100 days after transplant, two stool samples will be collected at regularly scheduled follow up appointments (near day 60 and day 100). No product (inulin or placebo) will be given during this time frame. The study period ends 100 days after transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Age 2-18 years
2. Allogeneic Stem Cell transplant
3. Myeloablative therapy
4. Inpatient at Lurie Children's Hospital

Exclusion Criteria:

1. Previous Hematopoietic Stem Cell Transplant
2. Autologous Stem Cell Transplant
3. Reduced Intensity Conditioning used for transplant
4. History of ulcerative colitis, Crohn's disease, irritable bowel syndrome, celiac disease
5. History of Type 1 or Type 2 Diabetes Mellitus
6. Previous abdominal surgery necessitating the use of an ostomy
7. G-tube dependence
8. Nasal gastric/oral gastric tube dependence prior to starting the conditioning process
9. Graft vs host disease prior to enrollment at any site
10. Children under 2 years of age - literature shows that the microbiome is still developing in children under two years of age, and this development may skew results

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
Change in alpha and beta bacterial diversity measures in stool | Change of baseline alpha and beta bacterial diversity at 100 days after transplant
  Compare the effect of oral inulin vs. placebo on alpha and beta bacterial diversity in the stool of children undergoing hematopoietic stem cell transplant
Change in Short Chain Fatty Acid (SCFA) levels in stool | Change in baseline SCFA levels in stool at 100 days after transplant
  Compare the effect of oral inulin vs. placebo on SCFA levels in the stool of children undergoing hematopoietic stem cell transplant

SECONDARY OUTCOMES:
Bacterial Resistance genes in stool | Measured at enrollment, on the day of transplant, 30 days after transplant, and near 100 days after transplant
  Determine the impact of inulin intake vs. placebo on the prevalence of genes associated with antibiotic resistance of children undergoing hematopoietic stem cell transplant

CONTACTS AND LOCATIONS:
Overall Officials: Mehreen M Arshad, MD, Principal Investigator — Lurie Children's/Northwestern
Locations (1):
- Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No